CLINICAL TRIAL: NCT01608126
Title: A Comparison of Medial Cervical Plexus Block Versus Combined (Superficial and Deep) Cervical Plexus Block for Carotid Endarterectomy: A Prospective, Randomized Single Blind Study
Brief Title: Medial Cervical Block for Carotid Endarterectomy Comparison With Standard Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Nalos MD (Other)
Responsible Party: Sponsor-Investigator, Daniel Nalos MD, Prim Daniel Nalos, MUDr., Head of Dept., Anaesthesiology and Critical Care, Masaryk Hospital Krajská zdravotní a.s.
Organization: Masaryk Hospital Krajská zdravotní a.s. (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Medial block II /nalos
Record Dates: First submitted 2012-05-25; First posted 2012-05-30 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Cervical Plexus Block Comparison
Keywords: Ultrasound; Cervical Plexus; Anesthesia, Conduction; Surgical Procedures, Elective; Atherectomy
MeSH Terms: interventions — Cervical Plexus Block

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combined Cervical Block (Active Comparator)
  Interventions: Procedure: cervical block
- Median Cervical Block US guided (Active Comparator)
  Interventions: Procedure: cervical block

INTERVENTIONS:
Procedure: cervical block — In brief, the superficial block was performed using a 22G needle (07 x 40 mm). The mixture injected was 15 ml of 0.5% bupivacaine + 10 ml of 1% lidocaine. Deep cervical plexus block was performed using a Stimuplex DR stimulating needle and the dose of anaesthetic used was 10 ml 0.5% bupivacaine + 5 ml 1% lidocaine applied in the vicinity of the C3 nerve root.
  The MCPB performed using ultrasound-guidance aiming specifically for the interfascia space. Eighteen ml of 0.375% bupivacaine was injected into the interfascia space at the level of C3 vertebral body using a 22G needle (07 x 40 mm).

SUMMARY:
The purpose of the study is to compare efficacy, complications and safety of the standard method of Combined (superficial and deep) cervical plexus block (SDCPB) with Ultrasound guided Medial Cervical plexus block technique (MCPB).

Hypothesis: Ultrasound assisted MCPB is safer than SDCPB with similar efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Elective Carotid Endarterectomy

Exclusion Criteria:

* Denied consent to block performance, Emergency procedure

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
number of additional applications of short-acting local anaesthetic | intraoperatively
  The number of times a surgeon would have to supplement the Regional Block with intrafield application of increments of short-acting local anaesthetic
patient satisfaction | 24 h after operation
Complications | perioperative

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Nalos, MUDr., Study Chair — Masaryk Hospital; Jiří Cihlář, Prof Ing, Principal Investigator — Purkynje University Ústí nad Labem; Luděk Vašátko, MUDr., Principal Investigator — Masaryk Hospital; David Bejšovec, MUDr., Principal Investigator — Masaryk Hospital
Locations (1):
- Krajská zdravotní, a.s. - Masarykova nemocnice v Ústí nad Labem, o.z., Ústí nad Labem, Czechia

REFERENCES:
- [Background] Pandit JJ, Satya-Krishna R, Gration P. Superficial or deep cervical plexus block for carotid endarterectomy: a systematic review of complications. Br J Anaesth. 2007 Aug;99(2):159-69. doi: 10.1093/bja/aem160. Epub 2007 Jun 18. PMID 17576970
- [Background] Hakl M, Michalek P, Sevcik P, Pavlikova J, Stern M. Regional anaesthesia for carotid endarterectomy: an audit over 10 years. Br J Anaesth. 2007 Sep;99(3):415-20. doi: 10.1093/bja/aem171. Epub 2007 Jul 9. PMID 17621600
- [Background] Ramachandran SK, Picton P, Shanks A, Dorje P, Pandit JJ. Comparison of intermediate vs subcutaneous cervical plexus block for carotid endarterectomy. Br J Anaesth. 2011 Aug;107(2):157-63. doi: 10.1093/bja/aer118. Epub 2011 May 24. PMID 21613278
- See also: Related Info — http://www.prolekare.cz/anesteziologie-intenzivni-medicina-clanek/povrchovy-a-medialni-cervikalni-blok-mri-studie-35916?search=superficial+and+interfascial+cervical
- See also: Related Info — http://www.prolekare.cz/anesteziologie-intenzivni-medicina-clanek/fascialni-koncept-36901?search=fascie+brachi%C3%A1ln%C3%ADho+
- See also: Related Info — http://www.prolekare.cz/anesteziologie-intenzivni-medicina-clanek/fascie-brachialniho-plexu-32413?search=fascie+brachi%C3%A1ln%C3%ADho+
- See also: Related Info — http://www.prolekare.cz/prakticky-lekar-clanek/regionalni-a-celkova-anestezie-konkurence-nebo-kooperace-24648?search=
- See also: Related Info — http://www.prolekare.cz/anesteziologie-intenzivni-medicina-clanek/ultrazvukem-navadeny-medialni-cervikalni-blok-36873?search=Nalos